CLINICAL TRIAL: NCT00758472
Title: ReCap Total Hip Resurfacing Prospective Data Collection
Status: Terminated | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet U.K. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BMET UK 08
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hip Resurfacing
  Interventions: Device: ReCap Total Hip Resurfacing

INTERVENTIONS:
Device: ReCap Total Hip Resurfacing — ReCap Total Hip Resurfacing
  Other Names: RECAP

SUMMARY:
Prospective data collection on survivorship of ReCap Total Hip Resurfacing

DETAILED DESCRIPTION:
Detailed protocol not available

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hip joint arthritis

Exclusion criteria:

- less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suitable for Total Hip Resurfacing
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2005-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
survival rate | 10 yr

CONTACTS AND LOCATIONS:
Overall Officials: Evert Smith, MD, Principal Investigator — North Bristol NHS Trust
Locations (2):
- United Kingdom (2):
  - Southmead Hospital, Bristol
  - Robert Jones & Agnes Hunt Orthopaedic & District Hospital NHS Trust, Oswestry